CLINICAL TRIAL: NCT06508099
Title: Randomized Study of Vitamin A and D Prophylaxis Before Allogeneic Related and Unrelated Hematopoietic Stem Cell Transplantation
Brief Title: Vitamin A and D Supplementation in Allogeneic HCT
Acronym: VitaStem
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director of RM Gorbacheva Research Institute, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/24-n
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Biphenotypic Acute Leukemia; Lymphoblastic Lymphoma; Chronic Myeloid Leukemia; Myelodysplastic Syndromes; Myeloprolipherative Neoplsm; Non-hodgkin Lymphoma
Keywords: allogeneic hematopoietic transplantation; vitamin A; vitamin D
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — Vitamin A; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin supplementation (Experimental): vitamin A 300 000 IU and vitamin D 100 000 IU on days -14 to -8 before transplantation
  Interventions: Drug: Vitamin A; Drug: Vitamin D3
- Routine care (No Intervention): Routine care

INTERVENTIONS:
Drug: Vitamin A — 300 000 IU single dose orally
  Arms: Vitamin supplementation
Drug: Vitamin D3 — 100 000 IU single dose orally
  Arms: Vitamin supplementation

SUMMARY:
The therapy under investigation is the addition of 300 000 IU of vitamin A and 100 000 IU of vitamin D before conditioning. The study will include patients with malignant diseases in hematologic response with indications for allogeneic transplantation with matched related or matched unrelated donor.

DETAILED DESCRIPTION:
Currently there is an emerging evidence of gut microbiota role in major complications of HCT, including GVHD, oral mucositis, infectious complications due to multi-drug resistant bacteria in the gut. Early exhaustion of most intestinal bacterial phyla after HSCT is documented in many studies. This effect of intensive anti-infectious therapy is well known. Most authors explain the disruption of intestinal microbiota by massive antibiotic treatment in order to prevent infectious complications due to immune deficiency following HCT. Early decrease in anaerobic bacteria (phylum Firmicutes) is revealed in many studies, with subsequent recovery of these bacterial populations within next 2 months. This time dynamics is in accordance with reported data on depletion of certain anaerobic gut bacteria, e.g., Ruminococcus, Faecalibacterium spp., Roseburia, Blautia post-transplant, being associated with severe complications in HCT patients. These results are in accordance with severe posttransplant dysbiosis at different mucosal sites post-HCT, as shown elsewhere by routine bacteriology techniques. The metabolism of bacteria with positive effect on GVHD includes both vitamin D and vitamin A. It was demonstrated that Ruminococcus abundance is dependent on vitamin A and D intake. Another bacteria genera Faecalibacterium prausnitzii, which is also reported to produce butyrate and reduce GVHD is also dependent on abundance of vitamin A. The big phylum Firmicutes are also dependant on vitamin D and their abundance is reported to be associated with lower incidence of immune complications and suppression of antibiotic-resistant strains. To summarize the idea of the study is based on modulation of gut microbiota, which in term may result in lower incidence of GVHD and toxic complications of HCT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: acute myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome, chronic myeloproliferative disease, chronic myeloid leukemia, lymphoblastic lymphoma, myeloma
* Standard disease risk: less than 5% clonal blasts in the bone marrow and the absence of blast forms in the peripheral blood at the time of inclusion in the study or at least partial response for lymphoproliferative neoplasms.
* Related compatible donor 10/10 HLA-matched or unrelated compatible donor 9-10/10 HLA-matched
* Age ≥18 years
* Absence of severe concomitant somatic diseases

Exclusion Criteria:

* - Severe organ failure: creatinine more than 2 norms; ALT, AST more than 5 norms; bilirubin more than 1.5 normal;
* respiratory failure more than 1 degree. or oxygen dependence
* Unstable hemodynamics;
* Uncontrolled bacterial or fungal infection at the time of inclusion, despite adequate antibacterial or antifungal therapy (CRP>70 mg/l at the time of inclusion).
* Karnofsky index less than 70%
* Repeated allogeneic transplantation of hematopoietic cells;
* Creatinine clearance below 60ml/min/1.73m2;
* Severe cardiac pathology, including a decrease in ejection fraction less than <50%, unstable angina, exertional angina of III-IV functional class, heart failure of III-IV functional class, arrhythmia grade V according to Lawn
* Severe decrease in lung function, FEV1 <50% or DLCO<50% predicted
* Pregnancy
* Somatic or mental pathology that does not allow signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of gastrointestinal acute GVHD | 125 days
  Cumulative incidence of patients with acute GVHD II-IV grade, competing risk is death, relapse and primary graft failure

SECONDARY OUTCOMES:
Incidence of HSCT-associated adverse events | 125 days
  Toxicity assessment is based on presence of NCI CTC AE 5.0 event grades 3-5. Veno-occlusive disease incidence and severity assessment is based on EBMT criteria 2020. Transplant-associated microangiopathy incidence assessment is based on Harmonization criteria. All toxicity measurements will be aggregated as severity scores
Infectious complications | 125 days
  Incidence of infections, including analysis of severe bacterial, fungal and viral infections incidence
Overall survival | 2 years
  Kaplan-Meier estimate of either relapse, primary or secondary graft failure or death from all causes
Event-free survival | 2 years
  Kaplan-Meier estimate of either relapse, primary or secondary graft failure or death from all causes
Overall cumulative incidence of acute GVHD grade II-IV | 125 days
  Cumulative incidence of patients with acute GVHD II-IV grade, competing risk is death, relapse and primary graft failure
Incidence of moderate and severe chronic GVHD | 2 years
  Cumulative incidence of patients with moderate and severe chronic GVHD according to NIH 2015 criteria, competing risk is death, relapse and primary graft failure
Non-relapse mortality analysis | 2 years
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
GVHD-relapse-free survival analysis | 2 years
  Kaplan-Meier estimate of death, acute GVHD grade III-IV, severe chronic GVHD or relapse
Cumulative incidence of primary and secondary graft failure | 125 days
  Cumulative primary and secondary graft failure, competing risk is death and relapse

CONTACTS AND LOCATIONS:
Locations (1):
- RM Gorbacheva Research Institute, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Written study proposal to Pavlov University Ethical Committee.
Supporting Information: Study Protocol
URL: https://cloud.mail.ru/public/RSLN/ra5hVE4ZA